CLINICAL TRIAL: NCT04696744
Title: Prospective Study for the Prognostic and Predictive Role of Circulating Tumor Cells in Patients With Oropharyngeal Squamous Cell Carcinoma: CTCO (Circulating Tumor Cells in the Oropharynx)
Acronym: CTCO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0446
Record Dates: First submitted 2020-12-21; First posted 2021-01-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Circulating Tumor Cell; Oropharyngeal Cancer
Keywords: CTC; Oropharynx; HNSCC
MeSH Terms: conditions — Neoplastic Cells, Circulating; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTCO: adults with squamous cell carcinoma of the oropharynx with a curative aim
  Interventions: Biological: CTC detection

INTERVENTIONS:
Biological: CTC detection — The collection and analysis of CTCs will be carried out in the following 6 steps: A blood sample will be taken: a maximum volume of 30 ml on 3 x 10 ml BD Vacutainer® EDTA tubes is required for the study.
  CTCs will be enumerated and characterized by immunofluorescence after immunostaining with the following antibodies: anticytokeratin, anti-CD44, anti-N-cadherin and anti-PD-L1.
  • - Secondary criterion(s) : Different tumor and clinical parameters will be analysed to find a correlation with CTC detection Gene expression profiles will be analyzed using the RNAseq single-cell at different times: before treatment, at interim times, and in case of relapse in order to establish correlations between patients at high risk of relapse and their molecular profiles

SUMMARY:
Head and neck cancers (HNSCC) are primarily squamous cell cancers represented by tumors of the upper aerodigestive tract. Locally advanced stages (stages III and IV) account for 50 to 70% of all presentations. The three main risk factors are smoking, alcohol and oropharyngeal infection with human papilloma virus (HPV).

Apart from HPV status, there is no biomarker for the prognosis in HSNCC patients. Circulating Tumor Cells (CTCs) can provide "real-time" information on tumor behavior and are already used in various cancers (colon, lung). Their detection has limited sensitivity and biomarkers cannot be used for early diagnosis, but may be useful during follow-up to assess local, regional or metastatic early tumor recurrence.

By using blood samples at different times (at diagnosis, after initial treatment and during follow-up), we will be able to measure the variation in quantification and establish a predictive role of these CTCs for the response to treatment.

Our hypothesis is that CTCs may have a key role, in addition to clinical and radiological examination, in detecting early tumor relapse.

We believe that the joint consideration of clinical parameters, treatment strategy and quantification of CTCs could optimize patient follow-up and management.

The CTC extraction system, ClearCell® FX from Biolidics, is an automated microfluidic enrichment system. It has the advantage of recovering fully intact and viable CTCs from a standard blood sample. The gentle sorting principle allows to preserve cell integrity and thus the expression of surface antigens. The CTCs thus isolated can then be re-cultured or analyzed by immunostaining. This high-performance technique, in operation since December 2017 in the Biochemistry Department of Pr Claire Rodriguez-Lafrasse (HCL), has demonstrated its usefulness in lung cancer.

Transcriptomic analysis of CTCs can be performed at the scale of a cell after isolation of the CTCs. CTCs can then be sequenced in RNAseq either in bulk (pool of cells) or cell by cell on our Illumina (Nextseq) sequencer, in order to define the heterogeneity of the tumor. Transcriptome analysis then provides information on the state of the cell as to its position in the epithelio-mesenchymal transition thanks to a molecular signature by phenotype. A priori-free characterization is therefore possible thanks to the RNAseq single-cell. This highly sensitive and innovative technique will allow the study of the gene expression profile of CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Squamous cell carcinoma proven on biopsy
* Oropharyngeal location
* Curative treatment by Surgery followed by radiotherapy (chemotherapy) Or Radiochemotherapy Or Induction chemotherapy (+/- surgery) + radiotherapy
* Did not object to their participation in the study

Exclusion Criteria:

* Carcinoma of the nasopharynx, larynx, oral cavity or hypopharynx
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult subjects with squamous cell carcinoma of the oropharynx with a curative treatment scheduled
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
characterization of CTCs | Day 1
  The CTCs will be extracted using Biolidic's ClearCell automaton which uses a microfluidic technique.
  The CTCs will be enumerated and characterized in immunofluorescence after immunostaining with the following antibodies: anticytokeratin, anti-CD44, anti-N-cadherin and anti-PD-L1.
characterization of CTCs | Month 4
  The CTCs will be extracted using Biolidic's ClearCell automaton which uses a microfluidic technique.
  The CTCs will be enumerated and characterized in immunofluorescence after immunostaining with the following antibodies: anticytokeratin, anti-CD44, anti-N-cadherin and anti-PD-L1.
characterization of CTCs | Month 10
  The CTCs will be extracted using Biolidic's ClearCell automaton which uses a microfluidic technique.
  The CTCs will be enumerated and characterized in immunofluorescence after immunostaining with the following antibodies: anticytokeratin, anti-CD44, anti-N-cadherin and anti-PD-L1.
characterization of CTCs | Month 18
  The CTCs will be extracted using Biolidic's ClearCell automaton which uses a microfluidic technique.
  The CTCs will be enumerated and characterized in immunofluorescence after immunostaining with the following antibodies: anticytokeratin, anti-CD44, anti-N-cadherin and anti-PD-L1.

CONTACTS AND LOCATIONS:
Overall Officials: Philouze Pierre, Dr, Principal Investigator — Service ORL Chirurgie Cervico-faciale
Locations (1):
- Service ORL Chirurgie Cervico-faciale (Pr Philippe CERUSE), Lyon, France

IPD SHARING:
Plan to Share IPD: No